CLINICAL TRIAL: NCT06450990
Title: Efficacy, Safety, and Dose-response of a Live Biotherapeutic Product (BGY-1601-VT) as a First-line Monotherapy in Women With Acute Vaginal Infection: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy, Safety, and Dose-response of a Live Biotherapeutic Product in Women With Acute Vaginal Infection
Acronym: ELINA
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NEXBIOME THERAPEUTICS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGY-1601-VT-001
Record Dates: First submitted 2024-05-30; First posted 2024-06-10 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Bacterial Vaginosis; Vulvovaginal Candidiasis
Keywords: Vaginal infection; Bacterial Vaginosis (BV); Vulvovaginal Candidiasis (VVC); Anaerobic bacteria; Prevotella; Gardnerella vaginalis; Candida albicans; Acute Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal; Vaginitis

STUDY DESIGN:
Intervention Model Description: This clinical trial is an Interventional, phase I-II, randomized, double-blind, parallel assignment, placebo-controlled, multiple-dosing regimen. The hypothesis of the trial is the superiority of the active treatment (dose #1 and/or dose #2) versus the placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BGY-1601-VT #1 (Experimental): Arm 1: BGY-1601#1: one verum tablet at Day 0 (D0) and one placebo tablet at Day 2 (D2)
  Interventions: Drug: BGY-1601-VT; Other: PLACEBO
- BGY-1601-VT #2 (Experimental): BGY-1601#2: one verum tablet at D0 and one verum tablet at D2
  Interventions: Drug: BGY-1601-VT
- PLACEBO (Placebo Comparator): Placebo: one placebo tablet at D0 and one placebo tablet at D2
  Interventions: Other: PLACEBO

INTERVENTIONS:
Drug: BGY-1601-VT — Live biotherapeutic product. The active product ingredient of the Investigational Medicinal Product (IMP) is the bacterial strain Lacticaseibacillus rhamnosus Lcr35.
  Other Names: BGY-1601 vaginal tablet
  Arms: BGY-1601-VT #1; BGY-1601-VT #2
Other: PLACEBO — Placebo
  Other Names: Placebo vaginal tablet
  Arms: BGY-1601-VT #1; PLACEBO

SUMMARY:
The purpose of this clinical trial is to investigate the clinical efficacy and safety of a Live Biotherapeutic Product (BGY-1601-VT) intended as a first line of treatment in cases of acute vaginal infection without upfront microbiological confirmed diagnosis

ELIGIBILITY:
Inclusion Criteria:

* Post-menarche woman aged 18 to 50 years old (inclusive),
* With suspected Bacterial Vaginosis (BV) and/or Vulvovaginal Candidiasis (VVC), presenting symptoms of acute vaginal infection
* No clinically significant and relevant abnormalities of medical history (including mental disorders) or physical examination,
* Able and willing to participate to the trial by complying with the protocol procedures as evidenced by her dated and signed informed consent form,

Exclusion Criteria:

* Other already diagnosed or suspected infectious causes of bacterial vaginal infection (e.g., Trichomonas vaginalis, Chlamydia trachomatis, Neisseria gonorrhoeae) within 1 month
* Current herpes simplex flare-up in the genital area,
* Vulvar condyloma due to the human papilloma virus;
* Vulvar dermatoses (e.g.: psoriasis or lichenification);
* Clinical diagnosis of BV or VVC within 4 months;
* Treatment with any antibiotic or antifungal therapy (local or systemic) within 2 months, regardless of the indication;
* Treatment with any local treatment (probiotics, antiseptic, etc.) within 1 month, regardless of the indication;
* Participant using any intravaginal product (local contraceptive [spermicide, hormonal ring], moisturizer, tampon, intimate hygiene product, etc.);
* Participant with a chronic disease or condition or treatment known to impact the immune system, including auto-immune disease, diabetes, cancer, renal failure, etc.
* Pregnant or breastfeeding patient or intending to become pregnant within 1 month ahead, or having given birth within 3 months;
* Participant in perimenopause, i.e. aged 45 years or more, with irregular menstrual cycles that could lead to a suspicion of menopause;
* With a known or suspected food allergy or intolerance or hypersensitivity to any of the trial intervention ingredient;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Estimated)
Dates: Start 2024-07-08 (Estimated); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
To compare the efficacy of BGY-1601-VT, dosing regimen #1 versus placebo and dosing regimen #2 versus placebo, to treat acute vaginal infection | Visit 2 (V2) = 7 days
  Percentage of responders with clinical cure at Visit 2 (V2) without rescue therapy

SECONDARY OUTCOMES:
To compare the efficacy of BGY-1601-VT, dosing regimen #1 versus placebo, dosing regimen #2 versus placebo, and dosing regimen #1 versus dosing regimen #2, to treat acute vaginal infection | Visit 2 (7 days) and Visit 3 (28 days)
  Percentage of responders with clinical cure at each timepoints without rescue therapy Percentage of participants with improved symptoms at the timepoints
To assess the safety of BGY-1601-VT in dosing regimen #1 and dosing regimethe safety of placebo #2, and | V2 (7 days) and V3 (28 days)
  Adverse Events (AEs) reported
To compare the evolution of Lcr35 into the vaginal microbiome between dosing regimen #1 and dosing regimen #2. | Visit 2 (7 days) and Visit 3 (28 days)
  quantitative Polymerase Chain Reaction (qPCR) Lcr35 in the vaginal microbiota

IPD SHARING:
Plan to Share IPD: No